CLINICAL TRIAL: NCT00868556
Title: fMRI of the Brainstem in Migraine Sufferers and Controls. Does Iron Deposition Correlate With Progression of Disease?
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Stewart Tepper MD, PI, Cleveland Clinic Foundation
Other Study IDs: V81708; Merck Grant IISP 36047
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-03

CONDITIONS: Episodic Migraine; Chronic Daily Migraine
Keywords: fMRI scans; episodic migraine sufferers; chronic migraine sufferers; non migraine sufferers (controls)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 episodic migraine sufferers
- 2 chronic migraine sufferers
- 3 non migraine sufferers (controls)

SUMMARY:
This is a 2 visit research study for patients with or without a diagnosis of migraine. Participants will be administered informed consent, have a medical history taken and a physical examination performed, and complete 3 questionnaires at the first visit. The participants will have a functional MRI performed after completion of Visit 1. Study stipends will be given for each completed research visit.

The purpose of this study is to potentially identify risk factors and/or biomarkers (which are differences in the brain structures)by comparing the brain MRI scans of migraine sufferers to brain scans of control persons to attempt to identify migraine progression using the functional MRI scans.

DETAILED DESCRIPTION:
At Visit 1, patients in 3 diagnostic arms,(consisting of subjects with episodic migraine, chronic daily migraine or non-migraineurs/controls), of 11 subjects each, will be consented and then have a physical exam, medical history and current medication use documented. Each of these enrolled subjects will have a PRIME MD assessment administered, and will complete the MIDAS and ASC-12 questionnaires.

At Visit 2 these same subjects will have an fMRI performed.

Subjects will be greater than age 18, have the appropriate diagnoses, be able to be consented and not be pregnant or have an inability to have the fMRI performed (have implanted metal devices, have severe claustrophobia).

ELIGIBILITY:
Inclusion Criteria:

* adult episodic, chronic or non-migraine sufferers able to consent

Exclusion Criteria:

* contraindication to MRI such as severe claustrophobia and implanted devices such as neurostimulators, pacemakers, aneurysm clips, etc
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 11 episodic migraine sufferers, 11 chronic migraine sufferers, 11 non-migraine sufferers
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
assess anatomical changes with emphasis in iron deposition in brainstem structures of migraineurs and controls | within a month after consent is obtained

SECONDARY OUTCOMES:
correlate outcomes with headache surrogates (frequency, time since onset and age) | within one month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Tepper, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Wolff HG. Headache and Other Head Pain, New York: Oxford Univ Press; 1963
- [Background] Welch KM, Nagesh V, Aurora SK, Gelman N. Periaqueductal gray matter dysfunction in migraine: cause or the burden of illness? Headache. 2001 Jul-Aug;41(7):629-37. doi: 10.1046/j.1526-4610.2001.041007629.x. PMID 11554950
- [Background] Siberstein SD, Lipton RB, Solomon S, Mathew NT. Classification of daily and near-daily headaches: proposed revisions to the IHS criteria. Headache. 1994 Jan;34(1):1-7. doi: 10.1111/j.1526-4610.1994.hed3401001.x. PMID 8132434
- [Background] Silberstein SD, Lipton RB, Sliwinski M. Classification of daily and near-daily headaches: field trial of revised IHS criteria. Neurology. 1996 Oct;47(4):871-5. doi: 10.1212/wnl.47.4.871. PMID 8857711
- [Background] Bigal ME, Tepper SJ, Sheftell FD, Rapoport AM, Lipton RB. Field testing alternative criteria for chronic migraine. Cephalalgia. 2006 Apr;26(4):477-82. doi: 10.1111/j.1468-2982.2006.01128.x. PMID 16556250